CLINICAL TRIAL: NCT00168402
Title: A Study Using Botulinum Toxin Type A in Patients With Axillary Hyperhidrosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Therapeutic Area Head, Allergan, Inc
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 191622-046
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2011-05-30 (Estimated); Status verified 2011-05

CONDITIONS: Hyperhidrosis
Keywords: Axillary Hyperhidrosis
MeSH Terms: conditions — Hyperhidrosis | interventions — Botulinum Toxins, Type A

INTERVENTIONS:
Drug: Botulinum Toxin Type A

SUMMARY:
This is a three-year study in subjects with axillary hyperhidrosis involving injection of Botulinum Toxin Type A into the axilla to reduce sweating.

ELIGIBILITY:
Inclusion Criteria:

* Marked axillary hyperhidrosis

Exclusion Criteria:

* Previous use of botulinum toxin for hyperhidrosis

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 193 (Actual)
Dates: Start 2002-02; Primary Completion 2005-10 (Actual); Study Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
Subject's assessment of the severity of hyperhidrosis

SECONDARY OUTCOMES:
Measurement of axillary sweat production